CLINICAL TRIAL: NCT02179268
Title: International Committee of Medical Journal Editors
Brief Title: Antidepressants and Bone Mineral Density
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Yiming Wang, Department of Psychiatry, the Affiliated Hospital, Guiyang Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: [2012] NO31260237/C090103
Record Dates: First submitted 2014-06-19; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Bone Mineral Density Quantitative Trait Locus 7
Keywords: Antidepressants; bone mineral density; bone turnover markers
MeSH Terms: interventions — Sertraline; Citalopram; Dexetimide; Venlafaxine Hydrochloride; Reboxetine; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- sertraline & control (Active Comparator): sertraline 50-150mg tables for 1 year,Control (cognitive behavioral therapy by psychiatrists, 50min, every week for three months, every month, for nine months).
  Interventions: Drug: sertraline; Drug: citalopram; Drug: venlafaxine; Drug: reboxetine; Behavioral: control
- citalopram & Control (Active Comparator): citalopram 20-40mg tables by mouth every day for 1 year, Control (cognitive behavioral therapy by psychiatrists, 50min, every week for three months, every month, for nine months).
  Interventions: Drug: sertraline; Drug: citalopram; Drug: venlafaxine; Drug: reboxetine; Behavioral: control
- venlafaxine & control (Active Comparator): venlafaxine 75-100mg tables by mouth every day for 1 year, Control (cognitive behavioral therapy by psychiatrists, 50min, every week for three months, every month, for nine months).
  Interventions: Drug: sertraline; Drug: citalopram; Drug: venlafaxine; Drug: reboxetine; Behavioral: control
- reboxetine & control (Active Comparator): reboxetine 4-8mg tables by mouth every day for 1 year, Control (cognitive behavioral therapy by psychiatrists, 50min, every week for three months, every month, for nine months).
  Interventions: Drug: sertraline; Drug: citalopram; Drug: venlafaxine; Drug: reboxetine; Behavioral: control

INTERVENTIONS:
Drug: sertraline — 50mg, 50-150mg/d,qd for one year
  Other Names: Zoloff
Drug: citalopram — 20mg, 20-40mg/d,qd,for one year
  Other Names: Cipramil
Drug: venlafaxine — venlafaxine,25mg, 75-100mg/d, bid, for one year
  Other Names: Effexor
Drug: reboxetine — reboxetine,4mg, 4-8mg/d,qd for one year
  Other Names: Edronax
Behavioral: control — 50min, every week for three months, every month, for nine months
  Other Names: cognitive behavioral therapy

SUMMARY:
The aim of this five arm randomized trial was thus to compare selective serotonin reuptake inhibitor (SSRI)sertraline and citalopram to a dual reuptake inhibitor venlafaxine, a nor-adrenaline reuptake inhibitor reboxetine and a control group receiving placebo, with the primary endpoint being bone mineral density, and secondary endpoints being bone turnover markers.

DETAILED DESCRIPTION:
These results have overt clinical implications. They suggest a noxious effect, particularly of selective serotonin reuptake inhibitor (SSRI) antidepressants, on bone. Osteoporosis and fracture is overtly the problem of the elderly. However, the process of skeletal consolidation begins in childhood and the corresponding phase of demineralisation proceeds at a glacial pace and lasts throughout adulthood, as a consequence antidepressant therapy is likely to have a substantive impact on a phenomenon likely to manifest decades hence. It is known that numerically small changes in bone mineral density are associated with a substantial increase in fracture risk. Because the SSRIs have only been in widespread use for two decades, it is plausible that the consequences of this adverse effect are yet to emerge. These data consequently suggest a recalibration of the risk/benefit ratio of this class of agents and additionally beg the question of the potential role of screening for bone mineral density in this at-risk population group.

ELIGIBILITY:
Inclusion Criteria:

* Participants needed to have a primary diagnosis of depression with Zung Self Rated Depression Scale (SDS) > 53, and Hamilton Depression Scale (HAMD) ≥20.

Exclusion Criteria:

* The patients with hyperparathyroidism, myeloma or other disorders known to affect bone metabolism
* Use of estrogen
* Calcitonin drugs
* Previous antidepressant or other psychiatric drug use or prior treatment history

Ages: 20 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
bone mineral density (BMD) | Change from Baseline in bone mineral density at one year

CONTACTS AND LOCATIONS:
Overall Officials: yiming wang, Ph.D, Study Chair — World Health Organization